Title: Promoting Radon Testing via Smartphone App: A Clinical Trial in a High Radon State

Unique Protocol Identification Number: CTR radon DaCCoTA National Clinical Trial (NCT) Identified Number: NCT04980521

### UNIVERSITY OF NORTH DAKOTA

# **Institutional Review Board Informed Consent Statement**

Title of Project: Promoting Radon Testing via Smartphone App: A Clinical Trial in a High

**Radon State** 

**Principal Investigator:** Dr. Soojung Kim, (701) 777-2473, soojung.kim@und.edu

Co-Investigator(s): Dr. David Schmitz, (701) 777-3264, david.f.schmitz@und.edu; Dr. Gary

Schwartz, (701) 777-6598, gary.schwartz@und.edu; Dr. Marilyn Klug, (701) 777-

6770, marilyn.klug@und.edu

# **Purpose of the Study:**

The purpose of this research study is to compare the effectiveness of radon information delivered via the radon app vs. a traditional approach (printed brochure). The prevalence of exceptionally high levels of residential radon in ND, coupled with public's poor understanding of this hazard, is a critical public health problem.

### **Procedures to be followed:**

You will either receive instructions explaining how to login to the radon education app on your smartphone and use it for the next three months or the process by which you will receive a series of three printed brochures via postal mail in the next three months. Next, you will be asked to complete a short online survey, which will take about 20 minutes.

#### Risks:

There are no risks in participating in this research beyond those experienced in everyday life.

### **Benefits:**

You will not benefit from participation in this research, but we hope that the research will provide a better understanding of how to increase the public's radon awareness.

### **Duration:**

You will either have the app installed on your phone for three months or be informed to receive three printed brochures via postal mail (one per month), and complete the online survey questionnaire. Taken together, the initial session should take about 30 minutes.

## **Statement of Confidentiality:**

If you are asked to use the app, the app you install on your phone has data security as guaranteed by the app-developing company, Triad Interactive Media. If you are informed to receive three printed brochures via postal mail, the online survey questionnaire will ask you to provide your mailing address. In addition, the online survey questionnaire will ask for your full name and UND email address to keep track of your research participation record. However, your mailing address, name, and email address will not be attached to your survey responses. Therefore, your responses are recorded anonymously. If this research is published, no information that would identify you will be included since your name is in no way linked to your responses.

All survey responses that we receive will be treated confidentially and stored on a secure server. However, given that the surveys can be completed from any computer (e.g., personal, work, school), we are unable to guarantee the security of the computer on which you choose to enter your responses. As a participant in our study, we want you to be aware that certain "key logging" software programs exist that can be used to track or capture data that you enter and/or websites that you visit.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# **Right to Ask Questions:**

The researchers conducting this study are Drs. Soojung Kim, David Schmitz, Gary Schwartz, and Marilyn Klug. You may ask any questions you have now. If you later have questions, concerns, or complaints about the research please contact Dr. Soojung Kim at 701-777-2473 during the day.

If you have questions regarding your rights as a research subject, you may contact The University of North Dakota Institutional Review Board at (701) 777-4279 or <a href="UND.irb@UND.edu">UND.irb@UND.edu</a>. You may contact the UND IRB with problems, complaints, or concerns about the research. Please contact the UND IRB if you cannot reach research staff, or you wish to talk with someone who is an informed individual who is independent of the research team.

General information about being a research subject can be found on the Institutional Review Board website "Information for Research Participants" <a href="http://und.edu/research/resources/human-subjects/research-participants.html">http://und.edu/research/resources/human-subjects/research-participants.html</a>

## **Compensation:**

- If you are enrolled in COMM 110 class, you will receive 0.5 extra course credit point, which is equivalent to the half-hour research participation. If you complete the second and final session, you will receive additional 0.5 extra credit point.
- If you are enrolled in COMM 102 class, you will meet the half-hour research participation requirement for completing this first session. If you complete the second and final session, you will meet additional half-hour research participation requirement.
- In addition to extra credit or meeting the research requirement, you will receive \$10 gift card for this initial session. If you complete the second and final session, you will receive another \$15 gift card.

There is another option to participating to meet the one-hour research requirement for your COMM 102 class or receive one extra credit for your COMM 110 class. This option is to read an article related to this research and prepare a two-page reaction to it. The person in charge will provide the article.

You may withdraw from the study at any time without losing the course points assigned by your instructor. If you choose not to participate, please consult your course instructor on other methods to earn course points.

# **Voluntary Participation:**

You do not have to participate in this research. You can stop your participation at any time. You may refuse to participate or choose to discontinue participation at any time without losing any benefits to which you are otherwise entitled.

You do not have to answer any questions you do not want to answer.

You must be 18 years of age older to participate in this research study.

Completion and return of the online survey form implies that you have read the information in this form and consent to participate in the research.

Please keep this form for your records or future reference.

### UNIVERSITY OF NORTH DAKOTA

# **Institutional Review Board Informed Consent Statement**

Title of Project: Promoting Radon Testing via Smartphone App: A Clinical Trial in a High

**Radon State** 

**Principal Investigator:** Dr. Soojung Kim, (701) 777-2473, soojung.kim@und.edu

Co-Investigator(s): Dr. David Schmitz, (701) 777-3264, david.f.schmitz@und.edu; Dr. Gary

Schwartz, (701) 777-6598, gary.schwartz@und.edu; Dr. Marilyn Klug, (701) 777-

6770, marilyn.klug@und.edu

### **Purpose of the Study:**

The purpose of this research study is to compare the effectiveness of radon information delivered via the radon app vs. a traditional approach (printed brochure). The prevalence of exceptionally high levels of residential radon in ND, coupled with public's poor understanding of this hazard, is a critical public health problem.

### **Procedures to be followed:**

In this second and final session, you will be asked to take another short survey that should last about 20 minutes.

#### Risks:

There are no risks in participating in this research beyond those experienced in everyday life.

### **Benefits:**

You will not benefit from participation in this research, but we hope that the research will provide a better understanding of how to increase the public's radon awareness.

### **Duration:**

This second and final session should take about 20 minutes.

# **Statement of Confidentiality:**

The online survey questionnaire asks for your full name and UND email address to keep track of your research participation record. However, your name and email address will not be attached to your survey responses. Therefore, your responses are recorded anonymously. If this research is published, no information that would identify you will be included since your name is in no way linked to your responses.

All survey responses that we receive will be treated confidentially and stored on a secure server. However, given that the surveys can be completed from any computer (e.g., personal, work, school), we are unable to guarantee the security of the computer on which you choose to enter your responses. As a participant in our study, we want you to be aware that certain "key logging" software programs exist that can be used to track or capture data that you enter and/or websites that you visit.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## **Right to Ask Questions:**

The researchers conducting this study are Drs. Soojung Kim, David Schmitz, Gary Schwartz, and Marilyn Klug. You may ask any questions you have now. If you later have questions, concerns, or complaints about the research please contact Dr. Soojung Kim at 701-777-2473 during the day.

If you have questions regarding your rights as a research subject, you may contact The University of North Dakota Institutional Review Board at (701) 777-4279 or <a href="UND.irb@UND.edu">UND.irb@UND.edu</a>. You may contact the UND IRB with problems, complaints, or concerns about the research. Please contact the UND IRB if you cannot reach research staff, or you wish to talk with someone who is an informed individual who is independent of the research team.

General information about being a research subject can be found on the Institutional Review Board website "Information for Research Participants" <a href="http://und.edu/research/resources/human-subjects/research-participants.html">http://und.edu/research/resources/human-subjects/research-participants.html</a>

# **Compensation:**

- If you are enrolled in COMM 110 class, by completing this second and final session, you will receive additional 0.5 extra credit point.
- If you are enrolled in COMM 102 class, by completing this second and final session, you will meet additional half-hour research participation requirement.
- In addition to extra credit or meeting the research requirement, you will receive another \$15 gift card for this second and final session.

There is another option to participating to meet the one-hour research requirement for your COMM 103 class or receive one extra credit for your COMM 110 class. This option is to read an article related to this research and prepare a two-page reaction to it. The person in charge will provide the article.

You may withdraw from the study at any time without losing the course points assigned by your instructor. If you choose not to participate, please consult your course instructor on other methods to earn course points.

## **Voluntary Participation:**

You do not have to participate in this research. You can stop your participation at any time. You may refuse to participate or choose to discontinue participation at any time without losing any benefits to which you are otherwise entitled.

You do not have to answer any questions you do not want to answer.

You must be 18 years of age older to participate in this research study.

Completion and return of the online survey form implies that you have read the information in this form and consent to participate in the research.

Please keep this form for your records or future reference.